CLINICAL TRIAL: NCT06638593
Title: MIRRORS-FROZEN - a Pilot Randomised Controlled Trial (RCT) Comparing Open Vs Robotic Surgery in the Management of Women with Complex Pelvic Adnexal Masses ≤ 8cm.
Brief Title: MIRRORS-FROZEN - Comparing Open Vs Robotic Surgery in the Management of Women with Complex Pelvic Adnexal Masses ≤ 8cm.
Acronym: MIRRORS-FROZEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Radwa Hablase, Principal Investigator, Royal Surrey County Hospital NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24SURN279899
Record Dates: First submitted 2024-09-27; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Ovarian Cancer; Ovarian Mass; Ovarian Cysts; Fallopian Tube Neoplasms; Adnexal Carcinoma; Adnexal Cyst; Adnexal Masses
Keywords: Robotic; adnexal masses; Adnexal cysts
MeSH Terms: conditions — Ovarian Neoplasms; Ovarian Cysts; Fallopian Tube Neoplasms; Carcinoma, Skin Appendage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: MIRRORS-FROZEN Protocol. (Experimental): Initial laparoscopic phase and thorough inspection of the abdomino-pelvic cavity to determine the feasibility of proceeding robotically, followed by robotic excision of the mass(es) and its retrieval in a bag if deemed suitable to proceed robotically. The mass or cyst will be sent for frozen section to determine the extent of the surgery. The surgery will continue robotically, with conversion to laparotomy considered at any point at the discretion of the individual surgeon.
  Interventions: Procedure: MIRRORS-FROZEN Protocol.
- Arm 2 : Standard open surgery. (Active Comparator): A midline abdominal incision will be made from the outset, with intraoperative frozen section assessment to determine the extent of the surgery.
  Interventions: Procedure: Standard open surgery

INTERVENTIONS:
Procedure: MIRRORS-FROZEN Protocol. — Initial laparoscopic phase and thorough inspection of the abdomino-pelvic cavity to determine the feasibility of proceeding robotically, followed by robotic excision of the mass(es) and its retrieval in a bag if deemed suitable to proceed robotically. The mass or cyst will be sent for frozen section to determine the extent of the surgery. The surgery will continue robotically, with conversion to laparotomy considered at any point at the discretion of the individual surgeon.
  Arms: Arm 1: MIRRORS-FROZEN Protocol.
Procedure: Standard open surgery — A midline abdominal incision will be made from the outset, with intraoperative frozen section assessment to determine the extent of the surgery.
  Arms: Arm 2 : Standard open surgery.

SUMMARY:
Adnexal masses are growths that can form in the ovaries or fallopian tubes for different reasons, such as hormonal changes, infection, or cancer. These masses may cause pelvic discomfort, pain, constipation, or no symptoms at all. When adnexal masses are found on scans, they are described in a certain way to indicate if they could represent early-stage cancer, and the word "complex" is used to refer to these masses. Surgery is often recommended, where the mass is removed and examined under the microscope during surgery in a process called (frozen section analysis); to determine its true nature.

It is still difficult to confirm cancer before surgery, and many of these masses turn out to be benign (not cancerous) or borderline (slow-growing tumours). Currently, doctors use open surgery with a cut from at least the belly button to the pubic bone to remove these masses. Patients with a cancer diagnosis will then have more surgical steps including assessment and sampling of various areas inside the abdomen (known as staging surgery) to see how far the cancer has spread.

Recovery after open surgery can be long and painful, with a slow return to normal daily activities. The trial investigators know from practice that robotic surgery has replaced open surgery for most benign adnexal diseases and other types of women's cancers, such as womb cancer. Recovery is quicker, with less pain and blood loss, allowing for a faster return to daily activities.

This study, MIRRORS-FROZEN (pilot), compares robotic versus the standard open surgery in managing women with complex adnexal masses of eight centimetres or less. The hope is to decrease the need for open surgery in patients with benign or borderline disease and to assess if robotic surgery has similar, worse, or better outcomes for patients with cancer.

MIRRORS-FROZEN is funded by Intuitive Foundation and GRACE Charity. The investigators will establish the feasibility of conducting a large multicentre randomized controlled trial in the future comparing certain cancer outcomes between robotic and open surgery.

DETAILED DESCRIPTION:
Open surgical staging is the current standard practice in managing women with complex adnexal masses suspicious of cancer. The diagnostic dilemma of early-stage ovarian cancer often leads to overtreatment by laparotomy in a number of patients with benign or borderline pathology.

MIRRORS-FROZEN (pilot) is a feasibility study that aims to establish whether the MIRRORS-FROZEN protocol can operate successfully and whether patients are willing to be recruited and randomized to either of the trial arms. The pilot trial also examines the feasibility and appropriateness of collecting a number of surgical, oncological, and patient-reported outcomes. The aim is to provide proof of concept that a larger, adequately powered multi-centre RCT is feasible.

Patients referred to the MDT with complex adnexal pelvic mass(es) or cyst(s) will be identified through the MDT meeting and screened against the eligibility criteria. Complex adnexal pelvic masses are defined as O-RADS-3 and deemed high risk of cancer as per subjective expert opinion, or O-RADS-4, O-RADS-5, and masses with an IOTA ADNEX score of ≥ 10%. As per standard practice, all patients referred with suspicious pelvic mass(es) will undergo a staging CT scan, serving as the primary screening tool to determine suitability for MIRRORS-FROZEN (pilot). In situations where MRI has been performed as staging imaging, the diameter of the cyst(s) or mass(es) will be used. The largest diameter of the cyst(s) or mass(es) should be ≤ 8 cm. In cases of bilateral masses or cysts, the larger cyst will be used to determine suitability for inclusion in the trial.

Potential participants will then be contacted by the trial coordinator or an appropriately trained member of the trial team to introduce the trial and provide the participant information leaflet and study consent form, along with the contact details of the trial team, at least 24 hours before the standard preoperative clinic appointment. Those who express interest in participating will undergo a comprehensive consent process conducted by an adequately trained member of the trial team. Following the consent process, baseline data collection will take place along with the baseline trial questionnaires.

All eligible participants who have consented to participate in the trial will be randomized using an online randomization service, Sealed Envelope™. Randomization will be at a ratio of 2:1 (MIRRORS-Frozen vs. standard treatment), using a simple randomization algorithm carried out by the trial coordinator/PI or a designated member of the trial team. After randomization and theatre allocation, participants will be contacted by a member of the trial team to inform participants of their allocation. No blinding or masking of allocation will occur, as both the participant and surgeon need to be aware of the allocation. The trial coordinator/PI and statistician will not be blinded to the groups.

Participants randomized to the MIRRORS-FROZEN protocol will undergo an initial laparoscopic phase. A thorough inspection of the abdomino-pelvic cavity will be performed to determine the feasibility of proceeding robotically. In patients randomized to the robotic arm and deemed suitable to proceed, peritoneal fluid or washings will be retrieved, followed by robotic excision of the mass(es) and its retrieval in a bag. The choice of specimen retrieval method, whether through a wound protector ring or vaginally, is left to the discretion of the individual surgeon. Following retrieval of the mass(es), it will be sent for frozen section analysis as per standard pathology department practice to determine the extent of the surgery.

The surgery continues robotically; however, conversion to laparotomy can be considered at any point at the discretion of the individual surgeon, in the event of surgical difficulty where it is felt to be in the patient's best interest. For example, in situations of complex adhesions or to achieve intact removal of the cyst.

Participants randomized to the open arm will start with a midline abdominal incision from the outset, with intraoperative frozen section assessment.

Frozen section results will determine the extent of surgery in both the trial arms and the following surgical steps to be performed in both trial arms: For participants with benign pathology, the surgery may either end or proceed to completion hysterectomy and removal of the remaining tube(s) and ovary(ies), based on the patient's preference and agreed consent. For participants with borderline pathology, surgical staging will be performed and includes: peritoneal biopsies of normal surfaces, including from the undersurface of the right hemidiaphragm, bladder reflection, Pouch of Douglas, right and left paracolic gutters, and both pelvic sidewalls; infracolic omentectomy; hysterectomy and contralateral salpingo-oophorectomy unless preservation of fertility is desired; and appendicectomy for mucinous tumours.

If the mass is malignant, surgical staging should include: peritoneal biopsies of normal surfaces, including from the undersurface of the right hemidiaphragm, bladder reflection, Pouch of Douglas, right and left paracolic gutters, and both pelvic sidewalls (4-6 biopsies); supracolic omentectomy; retroperitoneal lymph node assessment of pelvic and para-aortic nodes, with removal of enlarged lymph nodes as a minimum (may be omitted in mucinous tumours); hysterectomy and contralateral salpingo-oophorectomy apart from cases of apparent Stage 1A disease where fertility preservation is desired; and appendicectomy if abnormal.

The trial participants will be followed up for six weeks, and patient-reported outcome questionnaires will be collected at trial-specified points. The trial questionnaires include The European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 and the ovarian cancer module (EORTC QLQ-OV28) complementing the EORTC QLQ-C30. The Hospital Anxiety and Depression Scale (HADS), consisting of 14 items, scored on a Likert scale and 11-point pain scale (0-10), will be used. The EQ5D-5L questionnaire will also be used to collect health economic data.

All the required trial data will be recorded directly on an e-Case Record Form (eCRF) using The Research Electronic Data Capture (REDCap). The collection of Patient Reported Outcomes (PROMs) will be carried out via emails, containing a link sent to the trial participants at specific trial points. All trial appointments will be tailored around the patient's routine hospital visits, negating the need for extra visits.

Anticipating a small standardized difference and aiming to achieve 80% power for the main trial, the investigators aim to recruit 40 women within a 24-month recruitment window. This sample size is pragmatically set to provide precision in estimating predefined feasibility criteria, such as the consent rate, ensuring timely recruitment. The key feasibility parameters will be assessed, offering foundational insights for the main trial.

ELIGIBILITY:
Inclusion Criteria:

* Complex adnexal Pelvic mass/es ≤8 cm with no malignant disease outside the adnexae on CT or MRI.
* Women aged ≥18 & ≤100 years old.
* Patients who had given their signed and written informed consent

Exclusion Criteria:

* Adnexal pelvic mass > 8 cm.
* Radiological or histological or cytological evidence of stage III or IV disease.
* Lack of capacity to understand and give informed consent.
* Patients not suitable for laparoscopic surgery, such as but not limited to those with severe aortic stenosis.
* Any patient randomized to either of the study arms and found to have disease which appears greater than stage 1 will be withdrawn from the trial and treated according to the national guidelines

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
1. Recruitment Rate | Through study completion, an average of 24-26 months
  Defined as the percentage of patients who consent to participate out of the total number of patients offered inclusion in the study.
2. Randomization acceptability | Through study completion, an average of 24-26 months
  Defined as the percentage of participants who withdrew consent specifically due to randomization allocation, out of the total number of participants who initially consented.
3. Response rate to the trial questionnaires | Through study completion, an average of 24-26 months
  Defined as the percentage of received responses out of the total number of responses sent at each assessment point defined by the trial protocol.

SECONDARY OUTCOMES:
Rate of intra-operative cyst rupture with spillage within the peritoneal cavity | Through study completion, an average of 24-26 months
  Defined as the percentage of cysts that rupture during surgery out of the total number of operations performed, both overall and within each treatment arm. At the beginning of surgery, the integrity of the cyst wall will be documented in both trial arms, accompanied by taking illustrative images. Before sending the cyst for frozen section analysis, a photographic image will be captured to confirm its wall status. Additionally, histological gross inspections conducted before frozen section analysis will be incorporated into both the frozen section results and the final histology report
Rate of Conversion to open surgery | Through study completion, an average of 24-26 months
  The percentage of patients converted to open surgery after being deemed suitable for Robotic Surgery following the initial diagnostic laparoscopy, out of the total number of surgeries that begin as robotic procedures. ( only for MIRRORS-FROZEN arm).
Blood Loss | Through study completion, an average of 24-26 months
  Blood Loss during surgery in millilitres - documented at the completion of the surgery in both arms - expressed as median and range.
Number of units of blood transfused | Through study completion, an average of 24-26 months
  Number of units of blood transfused ( intraoperatively & post operative) - documented on discharge for both trial arms - Expressed as median and range.
Intraoperative complications | Through study completion, an average of 24-26 months
  Documented at the completion of the surgery for each patient in both arms - Expressed as the overall complication rate (number of complications divided by the number of patients) and the rate of each specific observed complication.
Perioperative complications | Through study completion, an average of 24-26 months
  Perioperative Complications ( up to time of discharge from hospital) and post operative ( Up to six weeks - post surgery)- Expressed as the overall complication rate (number of complications divided by the number of patients) and the rate of each specific observed complication.- Post operative complications will be recorded and classified using Clavien-Dindo Classification.
Length of hospital stay | Through study completion, an average of 24-26 months
  Number of days in hospital following operation. Operation date=day 0. Documented on discharge for both trial arms - expressed as median and range.
Days of ITU admission | Through study completion, an average of 24-26 months
  Number of days from date of surgery to date suitable for stepdown care- Operation date=day - documented on discharge for both trial arms - expressed as median and range.
Days to chemotherapy if indicated | Through study completion, an average of 24-26 months
  Days from operation date. Operation date=day 0 - Expressed as median and range.
Readmission rates | Through out the study and up to six weeks post- surgery
  Reasons of readmission to be recorded - Expressed as the proportion of patients requiring readmission out of the total number of patients in each trial arm.
Cost of MIRRORS-FROZEN protocol vs standard open surgery. | Through out the study and up to six weeks post- surgery
  Cost comparison focusing on resources used in hospital (surgery, length of stay, readmissions, outpatients, A&E) and in the community post discharge (primary and community care). Contacts with services and professionals will be converted to costs using validated national tariffs and NHS Reference costs.
  The primary health-related outcome for the economic analysis will be EQ-5D-5L, completed by participants at baseline and at each assessment point. Responses will be used to estimate the patients; health related quality of life (utility level) at each time point. This will be done by scoring the EQ-5D 5L using a validated national tariff. The utility scores will be integrated over time to provide the Quality Adjusted Life Years (QALYs), accrued by each participant over the duration of the trial.
  A comparison of the difference in costs and difference in QALYs over the trial period will be conducted using appropriate statistical tests to assess significance.
Pain assessment | Through out the study and up to six weeks post- surgery
  Numeric rating scale (NRS11) 0 (no pain) - 10 (worst pain) At baseline and post-operatively; day 1, 3, 7, 10, 14, 21, 6 weeks.
Quality of Life following surgery (generic) | Through out the study and up to six weeks post- surgery
  The EQ-5D-5L (EuroQol 5-Dimension 5-Level) assesses health through five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels (no problems to extreme problems), and responses form a 5-digit code describing the patient's health state. Additionally, the EQ VAS (Visual Analogue Scale) records the patient's self-rated health on a vertical scale from 0 ('worst health') to 100 ('best health'), with higher scores indicating better health outcomes. Results expressed as QALY gain using EQ5D-5L At baseline and post-operatively; day 1, 3, 7, 10, 14,21,6 weeks.
Quality of Life following Surgery (cancer specific) | Through out the study and up to six weeks post- surgery
  Assessed using patient reported outcome measure (PROM) European Organisation for Research and Treatment of Cancer (EORTC) Validated quality of life questionnaire (QLQ) for ovarian cancer (QLQ-C30/QLQ-OV28). This validated questionnaire consists of the core module and its associated ovarian cancer specific module. Completed at baseline, day 3 post surgery, 3 and 6 weeks post-surgery. The QLQ-C30 (Quality of Life Questionnaire-Core 30) and QLQ-OV28 (Quality of Life Questionnaire-Ovarian Cancer 28) are tools used to assess the quality of life in cancer patients. Both scales score from 0 to 100. For functioning scales (e.g., physical, emotional functioning), higher scores indicate better outcomes. For symptom scales (e.g., pain, fatigue), higher scores represent worse symptoms or poorer outcomes.
Mental wellbeing | Through out the study and up to six weeks post- surgery
  Hospital anxiety and depression scale (HADS) A (Anxiety) and D (Depression) scores are calculated separately. 0-7 = Normal, 8-10 = Borderline, 11-21 = Abnormal (case) Completed at baseline, day 3 post surgery, 3- and 6-weeks post-surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Surrey County Hospital NHS Foundation Trust., Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated from this current study will be available upon request from Miss Rdawa Hablase (r.hablase@nhs.net) as raw anonymised data for up to 5 years following completion and publication of the study. Participants have given their consent for the information collected from this study to be used to support other research in the future and to be shared anonymously with other researchers.
Supporting Information: Study Protocol, ICF
Time Frame: Up to 5 years following completion and publication of the study
Access Criteria: The datasets generated from this current study will be available upon request from Miss Radwa Hablase (r.hablase@nhs.net) as raw anonymised data